CLINICAL TRIAL: NCT07152223
Title: A Single-center Clinical Study to Evaluate the Safety and Efficacy of CD19-BCMA CAR-T Cell Therapy for Connective Tissue Diseases
Brief Title: Clinical Study on the Safety and Efficacy of CD19-BCMA CAR-T Cell Therapy for Connective Tissue Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-25-003
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Connective Tissue Diseases
Keywords: Connective Tissue Diseases
MeSH Terms: conditions — Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): The dosage range of 1.0 × 10^6/kg (± 20%) to 3.0 × 10^6/kg (± 20%) of CAR-T cells, administered intravenously.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Eligible subjects who successfully passed screening will receive CAR-T cell infusion on Day 0 after lymphodepleting preconditioning chemotherapy.

SUMMARY:
This study is a single-arm, single-center Investigator-Initiated Trial (IIT) designed to evaluate the safety, pharmacokinetic profile, and preliminary efficacy of CD19-BCMA CAR-T cells in subjects diagnosed with connective tissue diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Good compliance: The patient or their guardian understands and voluntarily signs the informed consent form, and it is expected that all documents, procedures, follow-up examinations and treatments stipulated in the study can be completed.
2. Previously diagnosed with one of the following diseases and meeting the corresponding latest international classification/diagnostic criteria :

   1. Systemic lupus erythematosus (SLE);
   2. Rheumatoid arthritis (RA);
   3. Systemic scleroderma (SSc) ;
   4. Sjogren's Syndrome (SS);
   5. Polymyositis/dermatomyositis (PM/DM);
   6. Mixed connective tissue disease (MCTD).
3. Researchers determine that the disease is in an active stage;
4. At least one autoantibody is positive in the serum or plasma during the screening period;
5. Insufficient response, intolerance or recurrence to at least one standard treatment;
6. The pregnancy test of the female subjects was negative, and the subjects agreed to take effective contraceptive measures throughout the trial period.
7. The patient's major tissues and organs are functioning well.

Exclusion Criteria:

1. Intracranial hypertension or confusion;
2. Symptomatic heart failure or severe arrhythmia;
3. Respiratory failure;
4. Accompanied by other types of malignant tumors;
5. Diffuse vascular coagulation;
6. Serum creatinine and/or urea nitrogen ≥ 1.5 times the normal value;
7. Sepsis or other difficult-to-control infections;
8. Uncontrollable diabetes;
9. Severe mental disorder;
10. Cranial magnetic resonance imaging (MRI) examination revealed obvious lesions in the intracranial cavity.
11. WHO physical status classification ≥ level 3;
12. Organ transplant recipients;
13. Pregnant and lactating women;
14. HIV+，HBV，HCV，EBV，CMV.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety | Up to 2 years after CAR-T infusion
  Count the Incidence of adverse events

SECONDARY OUTCOMES:
Effectiveness evaluation | Up to 2 years after CAR-T infusion
  The response rate of the responder index of systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), systemic sclerosis (scleroderma SSc), Sjogren's Syndrome, polymyositis/dermatomyositis, and mixed connective tissue disease (MCTD), as well as the changes in scores compared with the baseline value
Pharmacokinetic parameters | Up to 2 years after CAR-T infusion
  The highest concentration of CAR-T cell expansion in peripheral blood after administration.
Pharmacodynamic parameters | Up to 2 years after CAR-T infusion
  The peak values of CAR-T-related cytokines, which include at least IL-6 and IFN-γ.

CONTACTS AND LOCATIONS:
Overall Officials: Yuelin He, Ph.D. degree, Principal Investigator — Dongguan Taixin Hospital; Lan He, Ph.D. degree, Principal Investigator — Dongguan Taixin Hospital
Locations (1):
- Dongguan Taixin Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No